CLINICAL TRIAL: NCT02073682
Title: A Phase 3b, Prospective, Randomized, Open-label, Blind Evaluator (PROBE) Study Evaluating the Efficacy and Safety of (LMW) Heparin/Edoxaban Versus Dalteparin in Venous Thromboembolism Associated With Cancer
Brief Title: Cancer Venous Thromboembolism (VTE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DU176b-D-U311; 2014-004708-30 (EudraCT Number)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-09

CONDITIONS: Venous Thromboembolism (VTE); Deep Vein Thrombosis (DVT); Pulmonary Embolism (PE); Cancer
Keywords: Active Cancer with Metastasis
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Neoplasms | interventions — edoxaban; Dalteparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Edoxaban group (Experimental): After 5 days of low molecular weight heparin (LMWH), patients receive edoxaban treatment daily - tablet for oral use
  Interventions: Drug: Edoxaban; Drug: Low molecular weight heparin
- Dalteparin group (Active Comparator): Participants receive Dalteparin treatment daily -solution for subcutaneous injection
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Edoxaban — After the 5 day treatment with LMWH, patients receive edoxaban 60 mg once daily (QD) as 2 × 30 mg tablets (or 1 x 30 mg tablet QD for patients requiring dose adjustment) for the remainder of the treatment period.
  Other Names: DU-176b
  Arms: Edoxaban group
Drug: Dalteparin — Dalteparin was administered via subcutaneous injection at a dose of 200 IU/kg (maximum daily dose 18,000 IU) for 30 days, and at a dose of 150 IU/kg from Day 31 to the end of treatment.
  Other Names: Active comparator
  Arms: Dalteparin group
Drug: Low molecular weight heparin — Therapeutic doses of subcutaneous LMWH were administered for at least 5 days (to patients in the edoxaban group); this 5-day period may have included the pre-randomization LMWH (if applicable). The choice of parenteral LMWH was up to the treating physician.
  Other Names: LMWH
  Arms: Edoxaban group

SUMMARY:
The primary objective is to demonstrate the non-inferiority of edoxaban (preceded by a short course of LMWH) compared with dalteparin for the prevention of the combined outcome of recurrent venous thromboembolism (VTE) or major bleeding in subjects with VTE associated with cancer during a 12-month study period. If non-inferiority is established, LMWH/edoxaban will be compared with dalteparin for superiority.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with age ≥ 18 years or the otherwise legal lower age according to the country of residence;
* Confirmed acute lower extremity proximal DVT or PE for which long term treatment with low molecular weight heparin (LMWH) is indicated;
* Cancer, other than basal-cell or squamous-cell carcinoma of the skin;
* Able to provide written informed consent.

Exclusion Criteria:

* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current (index) episode of DVT and/or PE;
* Treatment with therapeutic doses of an anticoagulant other than that used for pretreatment of the current (index) VTE episode prior to randomization;
* Active bleeding or high risk for bleeding contraindicating treatment with LMWH or edoxaban;
* Any other contraindication listed in the local labeling of dalteparin, enoxaparin, or edoxaban;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1046 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (9):
- United States (4):
  - Brandon, Florida
  - Jonesboro, Georgia
  - Detroit, Michigan
  - Norfolk, Virginia
- Leuven, Vlaams-Brabant, Belgium
- Saint-Etienne, France
- Debrecen, Hajdu-Bihar Megye, Hungary
- Varese, Italy
- Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Patell R, Hsu C, Shi M, Grosso MA, Duggal A, Buller HR, Raskob G, Zwicker JI. Impact of mild thrombocytopenia on bleeding and recurrent thrombosis in cancer. Haematologica. 2024 Jun 1;109(6):1849-1856. doi: 10.3324/haematol.2023.284192. PMID 37855029
- [Derived] Raskob GE, van Es N, Verhamme P, Carrier M, Di Nisio M, Garcia D, Grosso MA, Kakkar AK, Kovacs MJ, Mercuri MF, Meyer G, Segers A, Shi M, Wang TF, Yeo E, Zhang G, Zwicker JI, Weitz JI, Buller HR; Hokusai VTE Cancer Investigators. Edoxaban for the Treatment of Cancer-Associated Venous Thromboembolism. N Engl J Med. 2018 Feb 15;378(7):615-624. doi: 10.1056/NEJMoa1711948. Epub 2017 Dec 12. PMID 29231094
- [Derived] van Es N, Di Nisio M, Bleker SM, Segers A, Mercuri MF, Schwocho L, Kakkar A, Weitz JI, Beyer-Westendorf J, Boda Z, Carrier M, Chlumsky J, Decousus H, Garcia D, Gibbs H, Kamphuisen PW, Monreal M, Ockelford P, Pabinger I, Verhamme P, Grosso MA, Buller HR, Raskob GE. Edoxaban for treatment of venous thromboembolism in patients with cancer. Rationale and design of the Hokusai VTE-cancer study. Thromb Haemost. 2015 Nov 25;114(6):1268-76. doi: 10.1160/TH15-06-0452. Epub 2015 Aug 13. PMID 26271200

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1050 participants were randomized from 114 sites in Western Europe (31), Central Europe (11), South Europe (36), Australia/New Zealand (13) and North America (23)
Pre-assignment Details: Of 1050 participants randomized, 1046 took study drug and were included in the modified Intent to Treat (mITT) and Safety Analysis Sets
Groups:
- Edoxaban Group: After 5 days of low molecular weight heparin (LMWH), participants received edoxaban treatment daily
- Dalteparin Group: Participants received dalteparin daily
Period: Overall Study
Arm/Group | Edoxaban Group | Dalteparin Group
Started | 522 | 524
Completed (In reasons not completed, acronyms are used: Investigator Decision (ID) and Patient Decision (PD)) | 200 | 154
Not Completed | 322 | 370
Not completed — Low Creatinine Clearance | 1 | 2
Not completed — Death | 86 | 100
Not completed — Cancer Cured | 10 | 15
Not completed — ID: Patient Noncompliance | 1 | 2
Not completed — ID: Palliative Treatment Only | 10 | 7
Not completed — Prohibited Concomitant Medication Use | 0 | 1
Not completed — Platelet Count <50,000/mL | 1 | 2
Not completed — Surgery/Medical Procedure | 3 | 1
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Start of New Chemotherapy Regimen | 6 | 3
Not completed — Cancer Progression | 53 | 33
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 79 | 62
Not completed — No reason provided | 11 | 9
Not completed — PD: Inconvenience of Dosing | 21 | 78
Not completed — Lost to Follow-up | 1 | 1
Not completed — ID: Benefit/Risk Judgment | 32 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban Group | Dalteparin Group | Total
Number analyzed (Participants) | 522 | 524 | 1046
Age, Continuous [Median (Full Range); unit: years] | 66 [22 to 91] | 65 [21 to 89] | 65 [21 to 91]
Age, Customized [Count of Participants; unit: Participants]
  18-64 Years | 246 | 261 | 507
  65-84 Years | 267 | 254 | 521
  85 years and over | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 261 | 506
  Male | 277 | 263 | 540
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The number analyzed in rows differs from overall because information was not provided by some participants: 13 in the edoxaban group and 18 in the dalteparin group.
  Participants
    White: number analyzed (Participants) | 509 | 506 | 1015
    White | 453 | 427 | 880
    Black or African American: number analyzed (Participants) | 509 | 506 | 1015
    Black or African American | 17 | 21 | 38
    Asian: number analyzed (Participants) | 509 | 506 | 1015
    Asian | 6 | 13 | 19
    Native Hawaiian/Pacific Islander: number analyzed (Participants) | 509 | 506 | 1015
    Native Hawaiian/Pacific Islander | 0 | 1 | 1
    Other: number analyzed (Participants) | 509 | 506 | 1015
    Other | 33 | 44 | 77
Region of Enrollment [Number; unit: participants]
  Netherlands | 61 | 57 | 118
  Belgium | 22 | 19 | 41
  Hungary | 17 | 16 | 33
  United States | 104 | 103 | 207
  Italy | 45 | 45 | 90
  France | 58 | 64 | 122
  Austria | 13 | 15 | 28
  Germany | 30 | 29 | 59
  Czechia | 11 | 10 | 21
  Spain | 35 | 35 | 70
  Australia | 16 | 16 | 32
  New Zealand | 12 | 13 | 25
  Canada | 98 | 102 | 200
Type of Cancer [Count of Participants; unit: Participants]
  Solid Tumor | 465 | 467 | 932
  Haematological Malignancy | 56 | 55 | 111
  Solid Tumor and Haematological Malignancy | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adjudicated Recurrent Venous Thromboembolism (VTE) or Major Bleeding Event
Time Frame: 12 months
Population: modified Intent to Treat (mITT), equating to the Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Group | Dalteparin Group
Number analyzed (Participants) | 522 | 524
Participants | 67 | 71
Statistical Analysis 1: Comparison: Edoxaban Group vs Dalteparin Group; Test type: Non-Inferiority — Edoxaban Group was considered non-inferior to the Dalteparin Group if the upper limit of the 2-sided 95% confidence interval (CI) for the Hazard Ratio ([LMW] Edoxaban Group to Dalteparin Group) was less than 1.5; p = 0.0056, Cox proportional hazard; Cox Proportional Hazard = 0.97, 95% CI 2-sided [0.696 to 1.359]
Statistical Analysis 2: Comparison: Edoxaban Group vs Dalteparin Group; Test type: Superiority — The hazard ratio (HR), two-sided confidence interval (CI) and p-value are based on the Cox proportional hazard model including treatment and the two stratification factors as covariates: the dichotomized bleeding risk and the dichotomized dose-adjustment factor; p = 0.8712, Cox proportional hazard

2. Secondary Outcome: Number of Participants With Adjudicated Major Bleeding Events While on Treatment
Description: The primary safety endpoint was major bleeding events during the On-Treatment Study Period (defined as on-study drug or up to 3 days after the last dose of study drug).
Time Frame: 12 months
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Group | Dalteparin Group
Number analyzed (Participants) | 522 | 524
Participants | 32 | 16
Statistical Analysis 1: Comparison: Edoxaban Group vs Dalteparin Group; The HR, 2-sided CI and p-value are based on the Cox regression model with counting process approach for on-treatment including treatment and the 2 stratification factors as covariates: the dichotomized bleeding risk and the dichotomized dose-adjustment factor; Test type: Superiority; p = 0.0254, Regression, Cox; Hazard Ratio (HR) = 2.0, 95% CI 2-sided [1.089 to 3.657]

3. Secondary Outcome: Number of Participants With Recurrent Venous Thromboembolism (VTE) During the Overall Study Period
Time Frame: 12 months
Population: mITT (Safety Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Group | Dalteparin Group
Number analyzed (Participants) | 522 | 524
Participants | 41 | 59
Statistical Analysis 1: Comparison: Edoxaban Group vs Dalteparin Group; The HR, 2-sided CI, and p-value are based on the Cox proportional hazard model including treatment and the 2 stratification factors as covariates: the dichotomized bleeding risk and the dichotomized dose-adjustment factor; Test type: Superiority; p = 0.0931, Cox proportional hazard; Cox Proportional Hazard = 0.71, 95% CI 2-sided [0.476 to 1.059]

4. Secondary Outcome: Number of Participants With Recurrent Deep Vein Thrombosis (DVT) During the Overall Study Period
Time Frame: 12 months
Population: mITT (Safety Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Group | Dalteparin Group
Number analyzed (Participants) | 522 | 524
Participants | 19 | 35
Statistical Analysis 1: Comparison: Edoxaban Group vs Dalteparin Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0394, Cox proportional hazard; Cox Proportional Hazard = 0.56, 95% CI 2-sided [0.318 to 0.972]

5. Secondary Outcome: Number of Participants With Recurrent Non-Fatal Pulmonary Embolism (PE) During the Overall Study Period
Time Frame: 12 months
Population: mITT (Safety Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Group | Dalteparin Group
Number analyzed (Participants) | 522 | 524
Participants | 21 | 24
Statistical Analysis 1: Comparison: Edoxaban Group vs Dalteparin Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.7324, Cox proportional hazard; Cox Proportional Hazard = 0.90, 95% CI 2-sided [0.502 to 1.624]

6. Secondary Outcome: Number of Participants With VTE-Related Death
Time Frame: 12 months
Population: mITT (Safety Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Group | Dalteparin Group
Number analyzed (Participants) | 522 | 524
Participants | 6 | 4
Statistical Analysis 1: Comparison: Edoxaban Group vs Dalteparin Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4873, Cox proportional hazard; Cox Proportional Hazard = 1.56, 95% CI 2-sided [0.444 to 5.505]

7. Secondary Outcome: Number of Participants With Recurrent VTE, Major Bleed or All-Cause Death
Time Frame: 12 months
Population: mITT (Safety Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban Group | Dalteparin Group
Number analyzed (Participants) | 522 | 524
Participants | 235 | 228
Statistical Analysis 1: Comparison: Edoxaban Group vs Dalteparin Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4199, Cox proportional hazard; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.898 to 1.293]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Edoxaban Group | Dalteparin Group
All-Cause Mortality (participants affected / at risk) | 206/522 | 192/524
Serious Adverse Events (participants affected / at risk) | 276/522 | 251/524
Other Adverse Events (participants affected / at risk) | 75/522 | 67/524
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edoxaban Group (N=522) | Dalteparin Group (N=524)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac mass (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 (12) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melaena (Gastrointestinal disorders) | 4 (4) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (5) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (2)
Death (General disorders) | 4 (4) | 4 (4)
Disease progression (General disorders) | 4 (4) | 2 (2)
Euthanasia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (4) | 2 (2)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Meningococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 16 (17) | 13 (13)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 7 (7)
Septic shock (Infections and infestations) | 3 (3) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 3 (3)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Huerthle cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 6 (6)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 69 (69) | 67 (67)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (24) | 21 (21)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulvar cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 4 (4)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 3 (3)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 6 (6) | 4 (4)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (3) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (6) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 16 (17)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 13 (13) | 8 (8)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (2) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edoxaban Group (N=522) | Dalteparin Group (N=524)
Deep vein thrombosis (Vascular disorders) | 34 (40) | 37 (45)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 41 (44) | 30 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT02073682/Prot_SAP_000.pdf